CLINICAL TRIAL: NCT03181269
Title: Human Milk and Infant Intestinal Microbiome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Joann McDermid, Joann M. McDermid, MSc, PhD, RDN, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB# 19913
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Breast Feeding; Human Microbiome
MeSH Terms: conditions — Breast Feeding | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention education (Experimental): Participants will receive the intervention education and data recording package.
  Interventions: Other: Intervention education
- Placebo education (Placebo Comparator): Participants will receive the placebo educational and data recording package.
  Interventions: Other: Placebo Education

INTERVENTIONS:
Other: Intervention education — An education package that includes an enhanced emphasis on maternal-infant skin-to-skin contact and a detailed activity log for recording early post-partum care practices that includes specific skin-to-skin contact time and frequency goals.
  Arms: Intervention education
Other: Placebo Education — An education package that includes a basic emphasis on maternal-infant skin-to-skin contact, as well as other general post-partum care practices and a general early post-partum care practices log without specific skin-to-skin contact goals.
  Arms: Placebo education

SUMMARY:
This study will explore the effects of skin-to-skin contact (SSC) between mothers and their babies on the infant intestinal microbiome, the maternal skin microbiome and the breast milk microbiome. This will be accomplished by administering an intervention education session to one group and a placebo education session to the second group in order to influence the magnitude of total SSC defined by the frequency and duration of contact time between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled to deliver at the University of Virginia Health System
* Women 18 years or older and their newborn infant
* Stated intent to exclusively breastfeed for the duration of post-partum hospital admission
* To have physical custody of their child when they are discharged from the hospital

Exclusion Criteria:

* Maternal antibiotic use in the 3 months prior to delivery
* Consumption of alcohol in the 3 months prior to delivery
* Recreational drug use in the 3 months prior to delivery
* Serious gastrointestinal conditions requiring medical intervention or medication during pregnancy (e.g. Crohn's disease, ulcerative colitis, celiac disease, gastrointestinal infections)
* Serious health conditions that require medication during pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Skin-to-skin contact | Duration of hospital admission after delivery (2-3 days)
  Self-reported magnitude of maternal-infant skin-to-skin contact

SECONDARY OUTCOMES:
Maternal skin microbiome | Duration of hospital admission after delivery (2-3 days)
  Maternal breast area skin microbiome
Maternal breast milk microbiome | Duration of hospital admission after delivery (2-3 days)
  Maternal first and early milk microbiome
Infant intestinal microbiome | Duration of hospital admission after delivery (2-3 days)
  Infant fecal microbiome
Maternal dietary intake | During pregnancy
  Maternal dietary intake of probiotic or culture-enhanced foods

CONTACTS AND LOCATIONS:
Overall Officials: Joann M McDermid, MSc PhD RDN, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pannaraj PS, Li F, Cerini C, Bender JM, Yang S, Rollie A, Adisetiyo H, Zabih S, Lincez PJ, Bittinger K, Bailey A, Bushman FD, Sleasman JW, Aldrovandi GM. Association Between Breast Milk Bacterial Communities and Establishment and Development of the Infant Gut Microbiome. JAMA Pediatr. 2017 Jul 1;171(7):647-654. doi: 10.1001/jamapediatrics.2017.0378. PMID 28492938
- [Background] Murphy K, Curley D, O'Callaghan TF, O'Shea CA, Dempsey EM, O'Toole PW, Ross RP, Ryan CA, Stanton C. The Composition of Human Milk and Infant Faecal Microbiota Over the First Three Months of Life: A Pilot Study. Sci Rep. 2017 Jan 17;7:40597. doi: 10.1038/srep40597. PMID 28094284
- [Background] Posthuma S, Korteweg FJ, van der Ploeg JM, de Boer HD, Buiter HD, van der Ham DP. Risks and benefits of the skin-to-skin cesarean section - a retrospective cohort study. J Matern Fetal Neonatal Med. 2017 Jan;30(2):159-163. doi: 10.3109/14767058.2016.1163683. Epub 2016 Mar 29. PMID 26955857
- [Background] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Background] Rutten N, Van der Gugten A, Uiterwaal C, Vlieger A, Rijkers G, Van der Ent K. Maternal use of probiotics during pregnancy and effects on their offspring's health in an unselected population. Eur J Pediatr. 2016 Feb;175(2):229-35. doi: 10.1007/s00431-015-2618-1. Epub 2015 Aug 30. PMID 26319129
- [Background] Jost T, Lacroix C, Braegger CP, Rochat F, Chassard C. Vertical mother-neonate transfer of maternal gut bacteria via breastfeeding. Environ Microbiol. 2014 Sep;16(9):2891-904. doi: 10.1111/1462-2920.12238. Epub 2013 Sep 3. PMID 24033881
- [Background] Schloss PD, Iverson KD, Petrosino JF, Schloss SJ. The dynamics of a family's gut microbiota reveal variations on a theme. Microbiome. 2014 Jul 21;2:25. doi: 10.1186/2049-2618-2-25. eCollection 2014. PMID 25061514
- [Background] Neu J, Rushing J. Cesarean versus vaginal delivery: long-term infant outcomes and the hygiene hypothesis. Clin Perinatol. 2011 Jun;38(2):321-31. doi: 10.1016/j.clp.2011.03.008. PMID 21645799
- [Background] Marin Gabriel MA, Llana Martin I, Lopez Escobar A, Fernandez Villalba E, Romero Blanco I, Touza Pol P. Randomized controlled trial of early skin-to-skin contact: effects on the mother and the newborn. Acta Paediatr. 2010 Nov;99(11):1630-4. doi: 10.1111/j.1651-2227.2009.01597.x. PMID 19912138
- [Background] Palmer C, Bik EM, DiGiulio DB, Relman DA, Brown PO. Development of the human infant intestinal microbiota. PLoS Biol. 2007 Jul;5(7):e177. doi: 10.1371/journal.pbio.0050177. Epub 2007 Jun 26. PMID 17594176
- [Background] Lindberg E, Adlerberth I, Hesselmar B, Saalman R, Strannegard IL, Aberg N, Wold AE. High rate of transfer of Staphylococcus aureus from parental skin to infant gut flora. J Clin Microbiol. 2004 Feb;42(2):530-4. doi: 10.1128/JCM.42.2.530-534.2004. PMID 14766812